CLINICAL TRIAL: NCT06034002
Title: A Phase 1, Open-Label, Multicenter Study of INCA033989 Administered as a Monotherapy or in Combination With Ruxolitinib in Participants With Myeloproliferative Neoplasms
Brief Title: A Study to Evaluate INCA033989 Administered as a Monotherapy or in Combination With Ruxolitinib in Participants With Myeloproliferative Neoplasms
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCA33989-102
Record Dates: First submitted 2023-08-30; First posted 2023-09-13 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Myeloproliferative Neoplasms
Keywords: Myeloproliferative Neoplasms; Myelofibrosis; Essential thrombocythemia; CALR mutation
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis; Thrombocythemia, Essential | interventions — ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1a Dose Escalation Cohort Disease Group A - with MF (Experimental): INCA033989 will be administered at a protocol defined starting regimen in 28-day cycles to identify the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE[s]). Participants with myelofibrosis (MF) will enroll in this group.
  Interventions: Drug: INCA033989
- Part 1a Dose Escalation Cohort Disease Group A - with ET (Experimental): INCA033989 will be administered at a protocol defined starting regimen in 28-day cycles to identify the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE[s]). Participants with essential thrombocythemia (ET) will enroll in this group.
  Interventions: Drug: INCA033989
- Part 1a: Dose Escalation Cohort Disease Group B - with TGB-MF SubOpt R (Experimental): INCA033989 will be administered at a protocol defined starting regimen in 28- day cycles and will allow for the evaluation of INCA033989 in combination with ruxolitinib to identify the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE[s]). Participants with myelofibrosis (MF) exhibiting suboptimal response (SubOpt R) will enroll in this group.
  Interventions: Drug: INCA033989; Drug: Ruxolitinib
- Part 1b: Dose Expansion - with MF (Experimental): INCA033989 will be administered as monotherapy at the RDE(s) identified during Part 1a. Participants with treatment group A (TGA) myelofibrosis MF will enroll in this group.
  Interventions: Drug: INCA033989
- Part 1b: Dose Expansion - with TGB-MF SubOpt R (Experimental): INCA033989 will be administered as an add-on therapy in combination with ruxolitinibat at the RDE(s) identified during Part 1a. Participants with treatment Group B (TGB) MF SubOpt R will enroll in this group.
  Interventions: Drug: INCA033989; Drug: Ruxolitinib
- Part 1b: Dose Expansion - with ET (Experimental): INCA033989 will be administered as monotherapy at the RDE(s) identified during Part 1a. Participants with treatment group A (TGA) essential thrombocythemia (ET) will enroll in this group.
  Interventions: Drug: INCA033989
- Part 1c: Dose Expansion (Experimental): INCA033989 will be administered at the dose level found to exhibit an overall positive benefit/risk as monotherapy or as combination therapy with Ruxolitinib. Participants with myelofibrosis (MF) will enroll in this group. The participants enrolled in the monotherapy arm will be offered the option to crossover to combination therapy with ruxolitinib if a suboptimal response to monotherapy is observed after 12 weeks.
  Interventions: Drug: INCA033989; Drug: Ruxolitinib

INTERVENTIONS:
Drug: INCA033989 — INCA033989 will be administered at protocol defined dose.
Drug: Ruxolitinib — Rux will be administered according to Prescribing Information/SmPC.
  Other Names: Jakafi
  Arms: Part 1a: Dose Escalation Cohort Disease Group B - with TGB-MF SubOpt R; Part 1b: Dose Expansion - with TGB-MF SubOpt R; Part 1c: Dose Expansion

SUMMARY:
This study is being conducted to evaluate the safety, tolerability, dose-limiting toxicity (DLT) and determine the maximum tolerated dose (MTD) and/or recommended dose(s) for expansion (RDE) of INCA033989 administered as a Monotherapy or in Combination With Ruxolitinib in participants with myeloproliferative neoplasms.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy > 6 months.
* Willingness to undergo a pretreatment and regular on-study BM biopsies and aspirates (as appropriate to disease).
* Existing documentation from a qualified local laboratory of CALR exon-9 mutation.
* Participants with MF or ET as defined in the protocol.

Exclusion Criteria:

* Presence of any hematological malignancy other than ET, PMF, or post-ET MF.
* Prior history of major bleeding, or thrombosis within the last 3 months prior to study enrollment.
* Participants with laboratory values exceeding the protocol defined thresholds.
* Has undergone any prior allogenic or autologous stem-cell transplantation or such transplantation is planned.
* Active invasive malignancy over the previous 2 years.
* History of clinically significant or uncontrolled cardiac disease.
* Active HBV/HCV or known history of HIV.
* Any prior chemotherapy, immunomodulatory drug therapy, immunosuppressive therapy, biological therapy, endocrine therapy, targeted therapy, antibody, or hypomethylating agent used to treat the participant's disease, with the exception of ruxolitinib for TGBs only, within 5 half-lives or 28 days (whichever is shorter) before the first dose of study treatment.
* Participants undergoing treatment with G-CSF, GM-CSF, or TPO-R agonists at any time within 4 weeks before the first dose of study treatment.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2028-10-29 (Estimated); Study Completion 2028-10-29 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities (DLTs) | Up to 28 days
  Dose-limiting toxicity will be defined as the occurrence of any of the toxicities as per protocol.
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 3 years and 60 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug, including those leading to dose modification or discontinuation.

SECONDARY OUTCOMES:
Participants with MF: Response using the revised IWG-MRT and ELN response criteria for MF | Up to 3 years and 60 days
  Defined as the percentage of participants with Response using the revised IWG-MRT and ELN response criteria.
Participants With MF: Percentage of participants achieving spleen volume reduction as defined in the protocol | Up to 24 weeks
  Defined as percentage of participants with a protocol defined Spleen Volume Reduction.
Participants with symptomatic anemia: Anemia Response as defined in the protocol | Up to 24 weeks
  Anemia Response as defined by the protocol.
Participants with ET: Response using the revised IWG-MRT and ELN response criteria for ET | Up to 3 years and 60 days
  Defined as the percentage of participants with Response using the revised IWG-MRT and ELN response criteria.
Incidence of AEs, ECGs, vital signs, and clinical laboratory evaluation | Up to 3 years and 60 days
  To evaluate the safety of INCA033989.
Percentage of participants achieving ≥ 50% reduction from baseline in total symptom score (TSS) | Week 12 and Week 24
  Defined as the percentage of participants achieving ≥ 50% reduction from baseline in TSS.
Mean change from baseline in TSS | Week 12 and Week 24
  Mean change in TSS from baseline.
Mean change in disease-related allele burden | Up to 3 years and 60 days
  Mean change from baseline in disease-related variant allele frequency quantified by targeted NGS and evaluated with myeloid and lymphoid proportion in blood.
Pharmacokinetics Parameter: Cmax of INCA33989 alone or for the combination of INCA033989 with ruxolitinib | Up to 3 years and 60 days
  Defined as maximum observed plasma concentration of INCA33989 alone or for the combination of INCA033989 with ruxolitinib.
Pharmacokinetics Parameter: Tmax of INCA033989 alone or for the combination of INCA033989 with ruxolitinib | Up to 3 years and 60 days
  Defined as the time to reach the maximum plasma concentration of INCA33989 alone or for the combination of INCA033989 with ruxolitinib.
Pharmacokinetics Parameter: Cmin of INCA33989 alone or for the combination of INCA033989 with ruxolitinib | Up to 3 years and 60 days
  Defined as the minimum observed plasma concentration of INCA33989 alone or for the combination of INCA033989 with ruxolitinib.
Pharmacokinetics Parameter: AUC(0-t) of INCA33989 alone or for the combination of INCA033989 with ruxolitinib | Up to 3 years and 60 days
  Defined as the area under the concentration-time curve up to the last measurable concentration of INCA33989 alone or for the combination of INCA033989 with ruxolitinib.
Pharmacokinetics Parameter: AUC 0-∞ of INCA33989 alone or for the combination of INCA033989 with ruxolitinib | Up to 3 years and 60 days
  Defined as the area under the concentration-time curve from 0 to infinity of INCA33989 alone or for the combination of INCA033989 with ruxolitinib.
Pharmacokinetics Parameter: CL/F of INCA33989 alone or for the combination of INCA033989 with ruxolitinib | Up to 3 years and 60 days
  Defined as the apparent oral dose clearance of INCA33989 alone or for the combination of INCA033989 with ruxolitinib.
Pharmacokinetics Parameter: Vz/F of INCA33989 alone or for the combination of INCA033989 with ruxolitinib | Up to 3 years and 60 days
  Defined as the apparent oral dose volume of distribution of INCA33989 alone or for the combination of INCA033989 with ruxolitinib.
Pharmacokinetics Parameter: t1/2 of INCA33989 alone or for the combination of INCA033989 with ruxolitinib | Up to 3 years and 60 days
  Defined as the apparent terminal phase disposition half-life of INCA33989 alone or for the combination of INCA033989 with ruxolitinib.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (13):
- United States (13):
  - City of Hope Medical Center, Duarte, California
  - Stanford Cancer Institute, Palo Alto, California
  - University of Miami Health System, Miami, Florida
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Icahn School of Medicine At Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Md Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A study to Evaluate INCA033989 Administered in Participants with Myeloproliferative Neoplasms — https://www.incyteclinicaltrials.com/study/?id=INCA33989-102&SearchTerm=INCA33989-102&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=